CLINICAL TRIAL: NCT05544916
Title: A Double-blind, Randomized, Placebo-controlled, Comparative, Multicenter Phase III Clinical Trial to Study the Clinical Efficacy and Safety of XC221, Tablets, 100 mg in Patients With Uncomplicated Influenza or Other Acute Respiratory Viral Infections
Brief Title: A Study to Evaluate the Safety and Efficacy of XC221 in Patients With Uncomplicated Influenza or Other Acute Viral Upper Respiratory Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XC221-03-04-2022
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Influenza; Respiratory Viral Infection
MeSH Terms: conditions — Influenza, Human | interventions — XC221

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XC221 (Experimental): Patients will take 1 tablet of XC221, tablets, 100 mg twice daily, in the morning (between 7:00 and 11:00 a.m.) and in the evening (between 7:00 and 11:00 p.m.), for 5 days.
  Interventions: Drug: XC221
- Placebo (Placebo Comparator): Patients will take 1 placebo pill orally twice a day, in the morning (between 7:00 and 11:00 a.m.) and in the evening (between 7:00 and 11:00 p.m.), for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC221 — 200 mg/day, for 5 days
  Arms: XC221
Drug: Placebo — 2 tablets/day, for 5 days
  Arms: Placebo

SUMMARY:
The main purpose of the study was to evaluate the effectiveness of XC221, tablets, at a dose of 200 mg/day compared to placebo in patients with uncomplicated influenza or other acute respiratory viral infections (ARIs).

An additional purpose of the study was to evaluate the safety of XC221, tablets, at a dose of 200 mg/day compared to placebo in patients with uncomplicated influenza or other ARIs.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 65 years inclusive;
2. Presence of written consent to participate in the study in accordance with applicable law;
3. Clinical signs of mild to moderate influenza or other acute respiratory infections (ARIs): an increase in body temperature, measured at the axilla, with a value between 38.0 °C and 39.5 °C, inclusive, during the current illness and without taking antipyretics within the last 8 h at the time of screening; at least one respiratory manifestation of influenza or other ARI (cough, runny nose/ stuffy nose, sore throat) of at least 2 points on a 4-point scale; at least one systemic manifestation of influenza or other ARI (headache, muscle pain, chills/sweating, fatigue) of at least 2 points on a 4-point scale.
4. No indication for hospitalization at the time of enrollment in the study;
5. Duration of illness from manifestation of symptoms to the first dose of study drug/placebo not more than 48 hours;
6. Negative pregnancy test for women of preserved reproductive potential;
7. Consent to use adequate contraceptive methods throughout the study and for 30 days after study completion;
8. Ability to understand the requirements for study participants, to give written consent to participate in the study (including the use and communication of patient health information relevant to the study) and to comply with the procedures of the study protocol.

Exclusion Criteria:

1. Pregnant and breastfeeding women;
2. Known hypersensitivity to the study drug, including the active and/or excipients.
3. Lactase deficiency, lactose intolerance, glucose-galactose malabsorption, galactose intolerance;
4. Diagnosis of COVID-19 established or probable at present (based on examination and analysis of epidemiological history);
5. Positive result of rapid test for SARS-CoV-2;
6. Blood oxygen saturation (SpO2) ≤ 95%, respiratory rate ≥ 22/min.
7. Complicated course of influenza or other acute respiratory infections;
8. Participation in any other clinical trial within 90 days prior to the screening period;
9. Known (based on medical history) or suspected alcohol abuse, psychotropic drugs, drug dependence, drug addiction;
10. Presence of mental illness, including a history of mental illness;
11. Clinical suspicion of pneumonia or other bacterial infections (including sinusitis, otitis media, urinary tract infection, meningitis, sepsis, etc.) requiring prescription of antibacterial drugs;
12. Taking antibiotics, antivirals, or immunomodulatory drugs for < 48 h before the study and/or plans to use these groups of drugs (other than the study drug) during the study;
13. Use of systemic, inhaled, or nasal glucocorticosteroids within 30 days prior to the study and/or plans to use glucocorticosteroids (except topical cutaneous agents) during the study;
14. Failure to withdraw for the duration of the study other medications that may affect the outcome of this study, such as antiviral medications, or medications that are incompatible with the study therapy;
15. Any cardiovascular, renal, hepatic, gastrointestinal, endocrine or nervous system diseases, severe decompensated chronic (including chronic kidney disease and chronic liver disease) or acute diseases or any other condition/disease that, in the opinion of the investigator, would make it unsafe for the patient to participate in the study;
16. Any vaccination of the patient within 90 days prior to inclusion in the study;
17. Diabetes mellitus in decompensation;
18. Obesity of 2-3 degrees (body mass index of 35 kg/m2 or more).
19. Patients who have undergone surgery within 30 days prior to the Screening Visit and patients who are scheduled to undergo surgery, including diagnostic procedures, or a hospital stay during the study;
20. The presence of cancer, including a history of cancer (with the exception of a cured tumor with sustained remission for more than 5 years);
21. The presence of HIV infection, tuberculosis, including in the anamnesis;
22. Meningeal syndrome;
23. Disturbance of consciousness (in the form of stunting, soporus, delirium, delirium, etc.).
24. Symptoms of pneumonia and possible acute respiratory distress syndrome (ARDS): cough with foaming sputum with blood, shortening of the pulmonary sound on percussion, a large number of different-caliber wet rales and abundant crepitation on auscultation, a sharp drop in blood pressure, deafness of heart tones and arrhythmia;
25. Patient's refusal to use approved contraception or to completely abstain from sexual intercourse for the duration of study participation, beginning at Visit 1, and for 30 days after completion of study participation;
26. Other reasons that, in the opinion of the investigator, prevent the patient from participating in the study or create an unreasonable risk.

Withdrawal Criteria:

1. Patient's desire to stop participating in the study (withdrawal of informed consent). Each patient has the right to stop participating in the study at any time without giving a reason. Withdrawal from the study will not affect the medical care provided to the patient in the future.
2. The decision by the research physician that the patient should be excluded is in the patient's own interest;
3. The need to prescribe etiotropic or any other treatment prohibited in the study, as determined by the investigating physician.
4. Patient refuses to cooperate with the investigator or is undisciplined;
5. Causes/occurrence during the study of situations that threaten patient safety (e.g., hypersensitivity reactions, serious adverse events, etc.);
6. Inclusion of a patient in the study with inclusion/inclusion criteria not met (prior to randomization);
7. Significant treatment failure; Significant failure is defined as a) skipping study drug/placebo for 2 consecutive days or more or b) taking, in total, < 80% or > 120% of the full course (full course = 10 pills).
8. Positive pregnancy test;
9. A confirmed diagnosis of COVID-19;
10. Occurrence in the course of the study of other reasons that prevent the study according to the protocol.
11. Death of a patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Time (in hours) from the first dose of the drug to the resolution of all of the ARI symptoms/events | Day 1 - Day 10
  Time (in hours) from the first dose of the drug to the resolution of all of the following symptoms/events.
  • fever (the day of fever resolution is the first day on which stable normal body temperature is achieved (<37.0°C without the use of antipyretics));
  All achieved symptoms/events scores maintained for at least 24 h at 0-1 point:
  * nasal congestion/runny nose;
  * sore throat;
  * cough;
  * muscle aches;
  * headaches;
  * fatigue;
  * chills/sweats. Patients will assess and record the severity of all symptoms on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.

SECONDARY OUTCOMES:
Time to decrease in 24-hour body temperature to ≤ 37.0°C without using antipyretics (number of hours from the first dose of the study treatment to a decrease in 24-hour body temperature to ≤ 37.0°C) | Day 1 - Day 10
  Patients will assess and record body temperature in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents
Time to nasal congestion/runny nose resolution (number of hours from the first dose of the drug to runny nose/congestion resolution, i.e. the time when the subject rates the 24-hour severity of this symptom at 0-1 point) | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom
Patient rate with reported nasal congestion/runny nose resolution by day 4 and day 6 from treatment initiation (i.e. patient rate who assessed the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Time to sore throat resolution (number of hours from the first dose of the drug to sore throat resolution, i.e. the time when the subject rates the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Patient rate with reported sore throat resolution by day 4 and day 6 from treatment initiation (i.e. patient rate who assessed the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 6
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Time to cough resolution (number of hours from the first dose of the drug to cough resolution, i.e. the time when the subject rates the 24-hour severity of this symptom at 0-1 point. | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Patient rate with reported cough resolution by day 4 and day 6 from treatment initiation (i.e. patient rate who assessed the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 6
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Time to muscle ache resolution (number of hours from the first dose of the drug to the resolution of muscle aches, i.e. the time when the subject rates the 24-hour severity of this symptom at 0-1 point | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Patient rate with reported muscle ache resolution by day 4 and day 6 from treatment initiation (i.e. patient rate who assessed the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 6
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Time to headache resolution (number of hours from the first dose of the drug to headache resolution, i.e. the time when the subject rates the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Patient rate with reported headache resolution by day 4 and day 6 from treatment initiation (i.e. patient rate who assessed the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 6
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Time to fatigue resolution (number of hours from the first dose of the drug to fatigue resolution, i.e. the time when the subject rates the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Patient rate with reported fatigue resolution by day 4 and day 6 from treatment initiation (i.e. patient rate who assessed the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 6
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Time to chills/sweats resolution (number of hours from the first dose of the drug to the resolution of chills/sweats, i.e. the time when the subject rates the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 10
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Patient rate with reported chills/sweats resolution by day 4 and day 6 from treatment initiation (i.e. patient rate who assessed the 24-hour severity of this symptom at 0-1 point). | Day 1 - Day 6
  Patients will assess and record the severity of symptom on a 4-point scale in the Patient's Diary for 10 days 2 times a day with a 12 ± 2 h interval before the next use of symptomatic agents, where: 0 points - no symptom; 1 point - the minimum severity of the symptom; 2 points - moderate severity of the symptom; 3 points - the maximum severity of the symptom.
Frequency complications of influenza or other viral upper respiratory tract infections (URIs) | Day 1 - Day 10
  Frequency complications of influenza or other viral URIs: sinusitis, otitis, bronchitis, pneumonia.
Time till elimination viruses based on qualitative polymerase chain reaction (PCR) test | Day 1 - Day 10
  Time to the first negative PCR test)
The need for paracetamol or ibuprofen: daily dose on days 1-10 | Day 1 - Day 10
  Dose of paracetamol or ibuprofen taken
Safety and Tolerability: adverse event (AE) rate | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 20 for each participant
  Number and frequency of adverse events (AEs) or serious AEs (SAEs)
Safety and Tolerability: AEs associated with the study drug | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 20 for each participant
  Number and frequency of AEs or SAEs) associated with the study drug
Safety and Tolerability: treatment discontinuation | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 20 for each participant
  Percentage of patients who discontinued treatment due to the occurrence of AEs/SAEs
Safety and Tolerability: hospitalization rate | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 20 for each participant
  Frequency of need for hospitalization due to AEs/SAEs
Safety and Tolerability: vital signs - systolic blood pressure (SBP) | Screening, day 4, day 6, day 10, and day 20 of the study or on the early termination visit, whichever came first, within 20 days of study participation
  SBP, mmHg
Safety and Tolerability: vital signs - diastolic blood pressure (DBP) | Screening, day 4, day 6, day 10, and day 20 of the study or on the early termination visit, whichever came first, within 20 days of study participation
  DBP, mmHg
Safety and Tolerability: vital signs - respiratory rate (RR) | Screening, day 4, day 6, day 10, and day 20 of the study or on the early termination visit, whichever came first, within 20 days of study participation
  RR, breaths per minute
Safety and Tolerability: vital signs - heart rate (HR) | Screening, day 4, day 6, day 10, and day 20 of the study or on the early termination visit, whichever came first, within 20 days of study participation
  HR, beats per minute
Safety and Tolerability: vital signs - body temperature | Screening, day 4, day 6, day 10, and day 20 of the study or on the early termination visit, whichever came first, within 20 days of study participation
  Body temperature, centigrade scale
Safety and Tolerability: physical examination results | Screening, day 4, day 6, day 10, and day 20 of the study or on the early termination visit, whichever came first, within 20 days of study participation
  Physical examination will follow the general rules of internal medicine: general examination, examination of mucous membranes and skin, including palpation of lymph nodes, evaluation of the musculoskeletal system, palpation, percussion, and auscultation of the main organ systems (cardiovascular, respiratory, digestive, and urinary systems) will be performed sequentially.
Safety and Tolerability: 12-lead electrocardiogram (ECG) - heart rate | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: heart rate (beats per minute)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - PQ interval | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: PQ interval (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - QRS complex | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QRS complex (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - corrected QT interval (QTc) | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QTc (ms)
Safety and Tolerability: complete blood count - hemoglobin | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Hemoglobin, g/dL
Safety and Tolerability: complete blood count - red blood cells | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Red blood cells, 10^6/uL
Safety and Tolerability: complete blood count - hematocrit | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Hematocrit, %
Safety and Tolerability: complete blood count - platelets | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Platelets, 10^3/uL
Safety and Tolerability: complete blood count - white blood cells | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  White blood cells, 10^3/uL
Safety and Tolerability: complete blood count - erythrocyte sedimentation rate | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Erythrocyte sedimentation rate, mm per hour
Safety and Tolerability: complete blood count - lymphocytes | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Lymphocytes, %
Safety and Tolerability: complete blood count - eosinophils | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Eosinophils, %
Safety and Tolerability: complete blood count - monocytes | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Monocytes, %
Safety and Tolerability: complete blood count - basophils | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Basophils, %
Safety and Tolerability: complete blood count - neutrophils | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Neutrophils, % (segmented and stab)
Safety and Tolerability: blood test results - glucose | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Glucose in blood serum, mmol/L
Safety and Tolerability: blood test results - total cholesterol | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Total cholesterol in blood serum, mmol/L
Safety and Tolerability: blood test results - triglycerides | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Triglycerides in blood serum, mmol/L
Safety and Tolerability: blood test results - total bilirubin | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Total bilirubin in blood serum, umol/L
Safety and Tolerability: blood test results - total protein | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Total protein in blood serum, g/L
Safety and Tolerability: blood test results - creatinine | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Creatinine in blood serum, umol/L
Safety and Tolerability: blood test results - urea | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Urea in blood serum, mmol/L
Safety and Tolerability: blood test results - aspartate transaminase (AST) | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  AST in blood serum, U/L
Safety and Tolerability: blood test results - alanine transaminase (ALT) | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  ALT in blood serum, U/L
Safety and Tolerability: blood test results - alkaline phosphatase (ALP) | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  ALP in blood serum, U/L
Safety and Tolerability: blood test results - creatine kinase (CK) | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  CK in blood serum, U/L
Safety and Tolerability: urinalysis - specific gravity | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Specific gravity of the urine
Safety and Tolerability: urinalysis - color | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Color of the urine
Safety and Tolerability: urinalysis - transparency | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Transparency of the urine
Safety and Tolerability: urinalysis - pH | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  pH of the urine
Safety and Tolerability: urinalysis - protein | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Protein in the urine (g/L)
Safety and Tolerability: urinalysis - glucose | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Glucose in the urine (mmol/L)
Safety and Tolerability: urinalysis (microscopy) - red blood cells | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Red blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - white blood cells | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  White blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - epithelial cells | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Epithelial cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - cylinders | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Cylinders in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - bacteria | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Bacteria in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - mucus | Screening, day 6, or on the early termination visit, whichever came first, within 20 days of study participation
  Presence of mucus in the urine

CONTACTS AND LOCATIONS:
Locations (13):
- Russia (13):
  - State autonomous health care institution "Engels City Clinical Hospital No. 1", Engel's
  - Medical Diagnostic Center "Medexpert", LLC, Engel's
  - Unimed-C Jsc, Moscow
  - Professors' Clinic LLC., Perm
  - Limited Liability Company "Health Energy", Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic No. 117", Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution "City polyclinic No. 112", Saint Petersburg
  - Limited Liability Company "Research Center Eco-Security", Saint Petersburg
  - Saint Petersburg State Budgetary Institution of Healthcare "City Pokrovskaya Hospital", Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic No. 4", Saint Petersburg
  - Limited Liability Company "Meili", Saint Petersburg
  - "Medical Clinic" Ltd., Saint Petersburg
  - State budgetary institution of health care of the Yaroslavl region "Clinical Hospital No. 2", Yaroslavl

IPD SHARING:
Plan to Share IPD: Undecided